CLINICAL TRIAL: NCT07183592
Title: Impact of Infusion Line Change Frequency on Infectious Complications Related to Central Venous Catheters in the Intensive Care Unit ICU
Brief Title: Impact of Infusion Line Change Frequency on Infectious Complications Related to Central Venous Catheters in the ICU - A Randomized Controlled Trial
Acronym: TANDOORI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 49RC24_0290; 2025-A01509-40 (Other: ANSM)
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Intensive Care (ICU); Central Venous Catheter Related Infections; Critical Care Nursing; Catheter-associated Bloodstream Infections (CLABSI); Nursing Workload

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7-day infusion set replacement (Experimental): Infusion sets connected to the central venous catheter will be replaced every 7 days.
  Interventions: Procedure: 7-day Infusion set replacement
- 4-day infusion set replacement (Active Comparator): Infusion sets connected to the central venous catheter will be replaced every 4 days.
  Interventions: Procedure: 4-day infusion set replacement

INTERVENTIONS:
Procedure: 7-day Infusion set replacement — 7-day infusion set replacement (Experimental arm) In this group, the infusion sets (the tubes and connectors used to deliver medications through the central venous catheter) will be changed once a week, every 7 days. During each replacement, all sets will be disconnected and replaced with new sterile ones.
  Arms: 7-day infusion set replacement
Procedure: 4-day infusion set replacement — 4-day infusion set replacement (Active comparator arm) In this group, the infusion sets will be changed every 4 days, which reflects the most common international recommendation. The procedure is the same: all sets connected to the central venous catheter will be replaced with new sterile ones. This strategy represents the current standard of care and will serve as the comparison for the 7-day approach.
  Arms: 4-day infusion set replacement

SUMMARY:
In the intensive care unit, patients' care and secure drugs administration require a central venous catheter. These invasive devices can lead to complications, particularly infections. Most preventive recommendations focus on catheter insertion, line handling, and dressings. Few recommendations adress catheter dwell time, which is certainly the main source of infection. Part of the prevention strategy is the regular and systematic replacement of infusion sets , as they may become contaminated during use, mainly through the hands of healthcare professionals. Prolonged use increases the risk of infection. Infusion lines changes involve disconnecting the old sets, discarding infusion devices containing drug residues, and replacing them with new sterile devices.

Current international guidelines recommend replacing these sets every 4 days, and the Center for Disease Control and Prevention recommends not exceeding 7 days. Replacing these devices requires the time of qualified nurses, numerous sterile medical devices, and medications. In addition to the intended effect on infection prevention, the procedure has impacts on workload and costs.

The objective of the study is to demonstrate that changing infusion set every 7 days does not increase the rate of central venous catheters related infections compared with changing infusion set every 4 days.

ELIGIBILITY:
Inclusion criteria

* Adult patient
* Any ICU patient with a central venous catheter (inserted by venipuncture) in place for less than 72 hours and with an expected dwell time of at least 7 days
* Patient affiliated with or covered by a social security system
* Patient who has given verbal consent or written consent from a third party or in the event that the patient is unable to give consent.

Exclusion Criteria

* Patient with a documented bloodstream infection at the time of inclusion
* Patient whose central venous catheter has been in place for more than 72 hours
* Patient with suspected catheter-related infection
* Patient whose study catheter was inserted using a guidewire exchange
* Patient previously enrolled in the study during the same ICU stay
* Patient whose condition, according to the clinician, does not allow safe placement of a central venous catheter, such as:

  * Allergy to catheter material
  * Confirmed deep vein thrombosis at the time of insertion
  * Inflammatory skin disorder at the insertion site
* Patient admitted for extensive burns
* Inadequate understanding of the French language
* Pregnant, breastfeeding, or postpartum woman
* Person deprived of liberty by judicial or administrative decision
* Person receiving involuntary psychiatric care
* Person under legal guardianship or other legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2830 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Rate (%) of patients with with a central venous catheter-related infectious complication | From central venous catheter insertion until 48 hours after catheter removal during the ICU stay (censored at 90 days).
  Infectious complications include:
  1. Catheter-related infections (CRI) defined as:
     * A positive catheter culture, with quantitative culture ≥10³ CFU/ml (Brun-Buisson technique) or, if not available, a semi-quantitative culture >15 CFU (Maki technique), and purulence at the catheter insertion site or tunnelitis.
     Or
     * A positive catheter culture, with quantitative culture ≥10³ CFU/ml (or semi-quantitative culture >15 CFU), and complete or partial regression of systemic signs of infection within 48 hours after catheter removal.
  2. Catheter-related bloodstream infections (bacteremia or fungemia) defined as:
     * The occurrence of bacteremia (or fungemia) within 48 hours before or after catheter removal (or suspected catheter-related infection if the catheter is not immediately removed), And
     * Either a positive culture with the same microorganism from the insertion site or catheter, with ≥10³ CFU/ml (Brun-Buisson technique) or, if not available, a semi-quantitative culture

SECONDARY OUTCOMES:
Central line-associated bloodstream infection (CLABSI) | Day 90
  Proportion of patients with central line-associated bloodstream infection
Non-central line-associated bloodstream infection | Day 90
  Proportion of patients with non-central line-associated bloodstream infection
Catheters with catheter colonization | From central venous catheter insertion until 48 hours after catheter removal during the ICU stay (censored at 90 days).
  Proportion of catheters with catheter colonization
Time to onset of central venous catheter-related infectious complication | Day 90
  Length of time (in days) before the onset of central venous catheter-related infectious complications
ICU length of stay | Day 90
  Length of ICU stay
All-cause ICU mortality | Day 90
  Number of patients who die from any cause during their ICU stay
Cumulative nursing time related to infusion set replacements | 1000 days
  Total nursing time, measured in minutes, required to perform infusion set replacements, per 1000 catheter-days
Cost of materials required for infusion set replacements | 1000 days
  Cost (euros) of materials required for infusion set replacements, per 1000 cathéter days

CONTACTS AND LOCATIONS:
Overall Officials: Carole Haubertin, Principal Investigator — University Hospital, Angers
Locations (20):
- France (20):
  - La Réunion University Hospital, Saint-Pierre, La Réunion
  - Albi Hospital, Albi
  - Angers University Hospital, Angers
  - Belfort Hospital, Belfort
  - Bourges Hospital, Bourges
  - Caen University Hospital, Caen
  - Chartres Hospital, Chartres
  - Cholet Hospital, Cholet
  - Colombes Hospital, Colombes
  - Corbeil-Essonnes Hospital, Corbeil-Essonnes
  - AP-HP - Henri Mondor Hospital, Créteil
  - Dijon University Hospital, Dijon
  - Garches Hospital, Garches
  - Le Puy en Velay Hospital, Le Puy-en-Velay
  - Macon Hospital, Mâcon
  - Nantes University Hospital, Nantes
  - Orleans University Hospital, Orléans
  - AP-HP - Tenon Hospital, Paris
  - Pontoise Hospital, Pontoise
  - Strasbourg University Hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided